CLINICAL TRIAL: NCT00839072
Title: Crossover Comparative Bioavailability Study of Trazodone Contramid(r) OAD 300 mg Extended-release Caplets and Desyrel(r) 100 mg Immediate-release Tablets in Healthy Adult Volunteers Under Fasting Conditions
Brief Title: Comparative Bioavailability Study of Extended-release and Immediate-release Trazodone in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Collaborators: Algorithme Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 04ACL1-011; TAN-P8-681
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Results first posted 2010-08-16 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: bioavailability; pharmacokinetics; healthy; crossover; trazodone
MeSH Terms: interventions — Trazodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trazodone Contramid OAD (Experimental)
  Interventions: Drug: Trazodone HCl
- Desyrel (Active Comparator)
  Interventions: Drug: Trazodone HCl

INTERVENTIONS:
Drug: Trazodone HCl — 100 mg immediate-release tablet, dosing q8h
  Arms: Desyrel
Drug: Trazodone HCl — 300 mg extended-release caplet, single dose
  Other Names: Oleptro
  Arms: Trazodone Contramid OAD

SUMMARY:
The objective of the study is to compare the pharmacokinetic profiles of extended-release and immediate-release trazodone formulations

DETAILED DESCRIPTION:
The bioavailability of once-daily trazodone extended-release 300 mg caplets (test product) and trazodone immediate-release 100 mg tablets administered q8h (reference product) will be compared in healthy adult volunteers in a randomized, crossover fashion. Morning doses will be administered after an overnight fast. Blood samples will be collected predose and at pre-defined times over 72 hours following the morning dose. Pharmacokinetic parameters will be analyzed using ANOVA. Comparative bioavailability will be assessed on the basis of the ratio of least-squares means and/or 90% confidence interval criteria.

ELIGIBILITY:
Inclusion Criteria:

* Availability for entire study period and willingness to adhere to protocol requirements as evidenced by signed informed consent
* Male or female volunteer, aged between 18 and 45 years inclusively
* BMI ≥20 and <30 kg/m2
* Minimum body weight: 60 kg
* Clinical laboratory values within normal range, or without clinical significance
* Healthy according to medical history, clinical laboratory results and physical examination
* Nonsmoker or ex-smoker

Exclusion Criteria:

* Significant history of hypersensitivity to trazodone or any related products, or severe hypersensitivity reactions to any drugs
* Presence or history of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs or known to potentiate or predispose to undesired effects
* Presence of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic, or dermatologic disease
* Suicidal tendency, history of or disposition to seizures, state of confusion, clinically relevant psychiatric disease
* Use of MAO inhibitors within 28 days of day 1 of the study
* Presence of significant heart disease or disorder according to ECG
* Seated systolic blood pressure lower than 90 or over 140 mmHg or diastolic blood pressure lower than 50 or over 90 mmHg at screening
* Maintenance therapy with any drug, or significant history of drug dependency or alcohol abuse (>3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Any clinically significant illness in the previous 28 days before day 1 of this study
* Use of any enzyme-modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem, and HIV antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, and rifampin), in the previous 28 days before day 1 of this study
* Females who are pregnant according to a positive serum pregnancy test, or are lactating
* Females of childbearing potential who refuse to use an acceptable method of contraception from the screening visit and throughout the study
* Volunteers who took an investigational product (in another clinical trial) or donated 50 mL or more of blood in the previous 28 days before day 1 of this study
* Poor motivation, intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with the protocol requirements or inability to cooperate adequately, inability to understand and to observe the instructions of the physician
* Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc) in the previous 56 days before day 1 of the study
* Positive urine screening for drugs of abuse
* Any history of tuberculosis and/or prophylaxis for tuberculosis
* Positive results to HIV, HBsAg, or anti-HCV tests

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-02; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma Inc., Laval, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Test (Trazodone Contramid® OAD) First: 1 * 300 mg Trazodone Contramid® OAD (Once-A-Day) Tablet Daily test product dosed in first period followed by Trazodone IR (Desyrel®) 100 mg tablet 8-hourly reference product dosed in the second period. The two periods were separated by a washout of at least 7 calendar days.
  IR = Immediate Release.
- Reference (Trazodone IR (Desyrel®) 100 mg 8-hourly) First: 1 * 100 mg Trazodone HCl IR (Desyrel®) Tablet 8-Hourly reference product dosed in first period followed by Trazodone Contramid® OAD (Once-A-Day) 300 mg Tablet Daily test product dosed in the second period. The two periods were separated by a washout of at least 7 calendar days.
  IR = Immediate Release.
Period: First Intervention Period
Arm/Group | Test (Trazodone Contramid® OAD) First | Reference (Trazodone IR (Desyrel®) 100 mg 8-hourly) First
Started | 12 | 12
Completed | 10 | 11
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 1
Period: Washout Period of 7 Days
Arm/Group | Test (Trazodone Contramid® OAD) First | Reference (Trazodone IR (Desyrel®) 100 mg 8-hourly) First
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | Test (Trazodone Contramid® OAD) First | Reference (Trazodone IR (Desyrel®) 100 mg 8-hourly) First
Started | 10 | 11
Completed | 9 | 11
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive Test first and Reference first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Region of Enrollment [Number; unit: participants]
  Canada | 24

OUTCOME MEASURES:

1. Primary Outcome: Bioequivalence Based on Cmax
Description: Cmax = Maximum plasma concentration Measured in nanograms per millilitre (ng/mL)
Time Frame: 72 hours post-dose
Population: The dataset for pharmacokinetic analysis comprised the 20 subjects who completed both study periods.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Trazodone Contramid® OAD: Trazodone Contramid® OAD 300 mg Tablets test product dosed in either period. In Period 1 subjects received either one tablet of the test formulation, Trazodone Contramid® OAD 300 mg, or three tablets 8 hours apart of the reference formulation, Desyrel® 100mg, after an overnight fast of at least 10 hours, followed by a 7 day washout period. In Period 2 subjects received the alternate regimen following an overnight fast of at least 10 hours.
  OAD = Once A Day
- Desyrel®: Desyrel® 100mg tablets reference product dosed in either period. In Period 1 subjects received either one tablet of the test formulation, Trazodone Contramid® OAD 300 mg, or three tablets 8 hours apart of the reference formulation, Desyrel® 100mg, after an overnight fast of at least 10 hours, followed by a 7 day washout period. In Period 2 subjects received the alternate regimen following an overnight fast of at least 10 hours.
  OAD = Once A Day
Arm/Group | Trazodone Contramid® OAD | Desyrel®
Number analyzed (Participants) | 20 | 20
ng/mL | 1060.8 (366.6) | 1743.3 (470.1)
Statistical Analysis 1: Comparison: Trazodone Contramid® OAD vs Desyrel®; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when the ratio of geometric Least Squares means (LS means) and confidence interval calculated from the exponential of the difference between the Test and Reference product for the ln-transformed parameter Cmax does not exceed 125%; Ratio of the mean = 59.66, 90% CI 2-sided [50.99 to 69.81] — Trazodone Contramid® OAD/Desyrel®

2. Primary Outcome: Bioequivalence Based on AUCT
Description: AUCT = Area under the concentration-time curve from 0 to the time of the last quantifiable concentration
Time Frame: 72 hours post-dose
Population: The dataset for pharmacokinetic analysis comprised the 20 subjects who completed both study periods.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Trazodone Contramid® OAD | Desyrel®
Number analyzed (Participants) | 20 | 20
ng*h/mL | 29180.6 (10557.1) | 36002.4 (9636.4)
Statistical Analysis 1: Comparison: Trazodone Contramid® OAD vs Desyrel®; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when the ratio of geometric Least Squares means and confidence interval calculated from the exponential of the difference between the Test and Reference product for the ln-transformed parameter AUCT is between 80% and 125%; Ratio of the mean = 78.55, 90% CI 2-sided [69.70 to 88.51] — Trazodone Contramid® OAD/Desyrel®

3. Primary Outcome: Bioequivalence Based on AUC∞
Description: AUC∞ = Area under the concentration-time curve extrapolated to infinity
Time Frame: 72 hours post-dose
Population: The dataset for pharmacokinetic analysis comprised the 20 subjects who completed both study periods.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Trazodone Contramid® OAD | Desyrel®
Number analyzed (Participants) | 20 | 20
ng*h/mL | 30913.7 (11904.8) | 37273.4 (10738.5)
Statistical Analysis 1: Comparison: Trazodone Contramid® OAD vs Desyrel®; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when the ratio of geometric Least Squares means and confidence interval calculated from the exponential of the difference between the Test and Reference product for the ln-transformed parameter AUC∞ is between 80% and 125%; Ratio of the mean = 80.05, 90% CI 2-sided [70.67 to 90.68] — Trazodone Contramid® OAD/Desyrel®

4. Secondary Outcome: Time of Maximum Measured Plasma Concentration (Tmax)
Time Frame: 72 hours post-dose
Population: The dataset for pharmacokinetic analysis comprised the 20 subjects who completed both study periods.
Measure: Median (Full Range); unit: hours
Arm/Group | Trazodone Contramid® OAD | Desyrel®
Number analyzed (Participants) | 20 | 20
hours | 6.00 [1.05 to 24.00] | 9.50 [0.33 to 21.00]

5. Secondary Outcome: Apparent Terminal Elimination Half-Life [T½el]
Description: The elimination half-life (T½el) of trazodone in plasma (time it takes for the concentration of trazodone to fall to half), expressed in hours.
Time Frame: 72 hours post-dose
Population: The dataset for pharmacokinetic analysis comprised the 20 subjects who completed both study periods.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Trazodone Contramid® OAD | Desyrel®
Number analyzed (Participants) | 20 | 20
Hours | 14.37 (4.31) | 12.16 (3.51)

6. Secondary Outcome: Area Under the Concentration-time Curve From 0 to 24 Hours [AUC0-24]
Time Frame: 24 hours
Population: The dataset for pharmacokinetic analysis comprised the 20 subjects who completed both study periods.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Trazodone Contramid® OAD | Desyrel®
Number analyzed (Participants) | 20 | 20
ng*h/mL | 16885.8 (5453.0) | 22512.8 (5045.2)

ADVERSE EVENTS:
Description: A total of 23 subjects were exposed to Trazodone Contramid® OAD during the study (12 during first intervention period and 11 during second intervention period).
  A total of 22 subjects were exposed to Trazodone IR (Apotex Corp.) during the study (12 during first intervention period and 10 during second intervention period).
Arm/Group | Trazodone Contramid® OAD | Desyrel®
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 20/23 | 21/22
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trazodone Contramid® OAD (N=23) | Desyrel® (N=22)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Dry eyes (Eye disorders) | 1 (1) | 2 (2)
Ocular hyperaemia (Eye disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 6 (9)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 6 (6) | 4 (5)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Hot flush (General disorders) | 1 (1) | 0 (0)
Vessel puncture site reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Blood potassium increased (Investigations) | 1 (1) | 1 (1)
Blood pressure systolic decreased (Investigations) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Nitrite urine present (Investigations) | 1 (1) | 1 (1)
Binocular eye movement disorder (Nervous system disorders) | 1 (1) | 0 (0)
Coordination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 9 (18)
Headache (Nervous system disorders) | 5 (6) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 17 (18) | 20 (39)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Approval from the sponsor will be required prior to publication of the results of this study and a draft manuscript will be submitted to the sponsor for scrutiny and comment. The choice of scientific journal will be mutually agreed on by the investigator and the sponsor.